CLINICAL TRIAL: NCT05134207
Title: The Effect of Oral Carbohydrate Solution Given Before Hip Artroplasty on Preoperative Anxiety and Postoperative Patient Comfort
Brief Title: The Effect of Oral Carbohydrate Solution on Anxiety and Comfort in Patients Undergoing Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevsehir Haci Bektas Veli University (Other)
Responsible Party: Principal Investigator, Gülden Küçükakça Çelik, assistant professor, Nevsehir Haci Bektas Veli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Record Dates: First submitted 2021-10-14; First posted 2021-11-24 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Hip Arthropathy; Fasting; Patient Comfort
Keywords: oral carbohydrate solution; anxiety; comfort
MeSH Terms: conditions — Fasting; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral carbohydrate solution (Experimental): Oral carbohydrate solution was given orally to the experimental group as 800 ml at 24:00 the night before the surgery and 400 ml at 06:00 2 hours before the intervention.
  Interventions: Dietary Supplement: oral carbohydrate solution
- control (No Intervention): From 24:00 on the night before the surgical intervention, food and water intake was prohibited for the patients in the control group.

INTERVENTIONS:
Dietary Supplement: oral carbohydrate solution — Patients in the intervention group; Preop oral carbohydrate solution was ingested orally twice within 10 minutes, as 800 ml at 24:00 the night before the surgery and 400 ml at 06:00 2 hours before the surgery.
  Arms: oral carbohydrate solution

SUMMARY:
Surgical interventions are not only a physiological trauma, but also a psychological and social trauma because they cause deterioration of the individual's comfort. Comfort is among the most basic human needs and provides a better care output. One of the conditions that cause deterioration of comfort and anxiety in patients is hunger and thirst before surgery. Since 1994, several guides published by professional groups in many countries on pre-operative fasting periods have published that clear liquids can be taken up to 2 hours before the surgery in elective surgeries, and solid foods can be taken up to 6 hours before the surgery. One of the basic principles of ERAS protocols, which include evidence-based care interventions applied at all stages of the surgical process, for the preoperative period is to ensure that the patient takes a carbohydrate drink up to two hours before anesthesia and to shorten the long fasting period. In many countries, the problems experienced by patients as a result of long-term hunger have been identified. When the comfort status of the patients who were given carbohydrate-rich drinks before the surgery was examined, it was observed that the symptoms such as thirst, hunger, insufficiency, fatigue, nausea, pain, anxiety and depression were reduced and oral carbohydrate solutions were recommended. In the literature, it is stated that the prolongation of the fasting period causes an increase in the anxiety of the person and negatively affects his comfort, and it is recommended to drink 800 ml of carbohydrate liquid food until midnight the day before the surgery and 400 ml of liquid carbohydrate food 2-3 hours before the surgery in order to provide metabolic satiety. The nurse, who is one of the health workers responsible for the care of the patient, has to manage the restriction of oral food and liquid intake and the comfort of the patient in the best way before the operation. Accordingly, in our study, the answers were sought whether the oral carbohydrate solution given before hip arthroplasty had an effect on anxiety and patient comfort.

DETAILED DESCRIPTION:
Hip arthroplasty (HA) is a very common treatment method in orthopedic surgery worldwide. HA is considered a successful, safe and cost-effective medical intervention to regain pain-free mobility and functionality of the hip joint in patients with severe joint disease or trauma.

It is stated that the annual number of patients undergoing HA in the United States is 193,000, and this number is approximately one million worldwide. In the next 15 years, it is estimated that the number of patients undergoing HA will continue to increase in the world and in Turkey.

It is stated that health care services should start in the preoperative period and continue in the postoperative period, especially in HA surgeries performed due to limitation of mobility. Because HA application is seen as a major surgical intervention and as with many surgical interventions, it can affect the individual as a whole.

Surgical intervention is a combination of anesthesia, drug therapy, tissue trauma, blood loss and body temperature changes. These developing events stimulate metabolic changes and cause postoperative anxiety and stress response at the same time. Exposure of the human body to surgery or other trauma elicits a neurohumoral response and activates a catabolic process. Surgical stress causes an increase in the release of regulatory hormones such as catecholamine, glucagon and cortisol in the body and a decrease in insulin sensitivity. The increase in cortisol level leads to the development of insulin resistance and hyperglycemia, which have an important effect on the healing process. Changes in this process increase the risk of postoperative complications and mortality.

On the other hand, fasting the patient overnight as a standard practice in the preoperative period in order to reduce the risk of lung aspiration in elective surgery patients may cause a change in the insulin glucagon ratio. This increases the stress response to surgical trauma and may have a major impact on glycemic control and insulin resistance. Prolongation of the preoperative fasting period may cause negative effects such as feeling of hunger, anxiety, restlessness, headache, dehydration, hypovolemia and hypoglycemia. However, the increase in the preoperative fasting period causes a decrease in patient satisfaction, and causes undesirable conditions such as nausea and vomiting in the postoperative period, delaying the healing process and prolonging the hospital stay of the patients.

In the guidelines published in countries such as America, Canada and Europe, it is reported that the longer the fasting period, the negative effects on patient safety and comfort. In elective surgeries, it is recommended that clear liquids can be consumed up to the last two hours and solid foods up to six hours before the surgical procedure in order to reduce anxiety, reduce the negative effects of the stress response on the patient, and ensure patient comfort. In the guideline published by the Turkish Society of Anesthesiology and Reanimation (TARD) in 2005, it is recommended to comply with these criteria in patients who will undergo elective surgery. Therefore, modern perioperative care aims at maximizing the shortening of the fasting period before an elective surgery.

According to Enhanced Recovery After Surgery (ERAS) protocols, one of the elements of modern perioperative care is the administration of preoperative oral carbohydrate loading (OCS). In the literature; oral carbohydrate solution administration before elective surgery; It is stated that it is absorbed from the stomach of the patient in an average of 90 minutes, reduces protein catabolism in the muscles, increases glycogen storage in the liver and reduces insulin resistance. In addition, in other studies conducted in abdominal, orthopedic and cardiac surgery; It has been determined that OCS reduces postoperative metabolic stress, preserves lean body mass and muscle strength, and increases patient comfort by reducing the length of hospital stay.

The concept of patient comfort is defined as the comfort that facilitates daily life. In providing the health care needs, which are extremely stressful for the patient, nurses apply nursing interventions for comfort, which is a concept unique to the individual, allowing the patient to experience less anxiety, be more peaceful and overcome their problems.

Discomforts experienced by the patient during the operation or procedures (pain, nausea, vomiting, hypothermia, anxiety, etc.) may increase the patient's anxiety and may be the main reason for the decrease in comfort. The nurse should provide all necessary nursing interventions to reduce or eliminate the situations that will cause anxiety in the patient before and after each procedure to be applied to the patient. With all these practices, patients can receive a quality nursing care, contribute to their faster recovery and increase their quality of life.

Quality patient care in surgical nursing; should be shaped within the framework of ethical principles such as not harming and providing benefit. In the literature; Evidence for the duration of fasting in the preoperative period is reflected in clinical practice, emphasizing the need to prevent patients from being harmed without putting them at risk. Thus, by managing the hunger period within the scope of evidence-based practices; It is stated that many therapeutic benefits can be obtained, such as reducing anxiety, discomfort, headache, thirst and hunger in the preoperative period, and providing patient comfort by reducing nausea, vomiting and dehydration in the postoperative period.

Managing food and fluid restriction in line with the guidelines in the preoperative period is one of the important responsibilities of the surgical nurse. Thus, the comfort of the patients will be increased, their anxiety will be reduced, and they will be able to return to their normal lives as soon as possible. Working from here; It was aimed to determine the effect of preoperative OCS on anxiety and patient comfort in patients undergoing HA.

ELIGIBILITY:
Inclusion Criteria:

* Who volunteered to participate in the research,
* Total hip replacement surgery planned,
* Who are over 18 years old,
* ASA I and II group,
* First time hip replacement surgery

Exclusion Criteria:

* Diabetes mellitus,
* In the emergency patient group,
* with gastroesophageal reflux,
* Those with esophageal disease (Hiatus hernia, esophagitis, achalasia…)
* Having endocrine problem,
* Diagnosed with ileus,
* With pyloric stenosis,
* ASA III and IV group,
* Intravenous fluid administered before surgery,
* Using drugs that affect blood glucose levels,
* Previous hip replacement surgery
* Body mass index over 35kg/m2 (The value obtained by dividing the weight in kilograms by the square of the height in meters),
* Having a psychiatric and neurological diagnosis, poor general condition,
* Needing all kinds of fluid and blood support in the pre-operative period,
* Patients who use alcohol or cigarettes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
preoperative anxiety | 10:00 pm the night before surgery
  State-Trait Anxiety Scale (The lowest score to be taken from the scale is 20, and the highest score is 80. High scores indicate high anxiety levels, low scores indicate low anxiety levels.
preoperative anxiety | just before the patient is sent for surgery
  State-Trait Anxiety Scale (The lowest score to be taken from the scale is 20, and the State-Trait Anxiety Scale (The lowest score to be taken from the scale is 20, and the highest score is 80. High scores indicate high anxiety levels, low scores indicate low
patient comfort | Considering that the discharge days of the patients would be different, it was applied on the second day after the operation.
  Post Hip Replacement Comfort Scale (The highest average score obtained from the scale is 5 and the lowest average score is 1. A high score indicates high comfort, and a low mean score indicates low comfort.)

SECONDARY OUTCOMES:
postoperative anxiety | Evaluated at 0th-hour, 2th-hour, 4th-hour, 6th-hour, 12th-hour postoperatively.
  Visual analog scale (Values range from 0 to 10 points, and higher values indicate increased severity of assessed symptoms.)
postoperative pain | Evaluated at 0th-hour, 2th-hour, 4th-hour, 6th-hour, 12th-hour postoperatively
  Visual analog scale (Values range from 0 to 10 points, and higher values indicate increased severity of assessed symptoms.)
postoperative sensation of thirst | Evaluated at 0th-hour, 2th-hour, 4th-hour, 6th-hour, 12th-hour postoperatively
  Visual analog scale (Values range from 0 to 10 points, and higher values indicate increased severity of assessed symptoms.)
postoperative nausea- vomiting | Evaluated at 0th-hour, 2th-hour, 4th-hour, 6th-hour, 12th-hour postoperatively
  Visual analog scale (Values range from 0 to 10 points, and higher values indicate increased severity of assessed symptoms.)
postoperative sensation of hunger | Evaluated at 0th-hour, 2th-hour, 4th-hour, 6th-hour, 12th-hour postoperatively
  Visual analog scale (Values range from 0 to 10 points, and higher values indicate increased severity of assessed symptoms.)
physiological parameter | preoperative night at 10 pm
  pulse rate/minute
physiological parameter | immediately before going to the operation
  pulse rate/minute
physiological parameter | postoperative 0th-hour, 2th-hour, 4th-hour, 6th-hour, 12th-hour.
  pulse rate/minute
physiological parameter | preoperative night at 10 pm
  respiratory rate/minute
physiological parameter | immediately before going to the operation
  respiratory rate/minute
physiological parameter | postoperative 0th-hour, 2th-hour, 4th-hour, 6th-hour, 12th-hour
  respiratory rate/minute
physiological parameter | preoperative night at 10 pm
  blood pressure (systolic and diastolic mmHg)
physiological parameter | immediately before going to the operation
  blood pressure (systolic and diastolic mmHg)
physiological parameter | postoperative 0th-hour, 2th-hour, 4th-hour, 6th-hour, 12th-hour
  blood pressure (systolic and diastolic mmHg)
physiological parameter | preoperative night at 10 pm
  oxygen saturation (SpO2, %)
physiological parameter | immediately before going to the operation
  oxygen saturation (SpO2, %)
physiological parameter | postoperative 0th-hour, 2th-hour, 4th-hour, 6th-hour, 12th-hour
  oxygen saturation (SpO2, %)
physiological parameter | preoperative night at 10 pm
  heat (Centigrade degree)
physiological parameter | immediately before going to the operation
  heat (Centigrade degree)
physiological parameter | postoperative 0th-hour, 2th-hour, 4th-hour, 6th-hour, 12th-hour
  heat (Centigrade degree)
physiological parameter | preoperative night at 10 pm
  blood glucose (mg/dL)
physiological parameter | immediately before going to the operation
  blood glucose (mg/dL)
physiological parameter | postoperative 0th-hour, 2th-hour, 4th-hour, 6th-hour, 12th-hour
  blood glucose (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Gülden Küçükakça Çelik, Phd, Principal Investigator — Nevşehir Hacı Bektaş Veli University
Locations (1):
- Gülden Küçükakça Çelik, Nevşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saray Kilic H, Tastan S. Development of post hip replacement comfort scale. Appl Nurs Res. 2017 Dec;38:169-174. doi: 10.1016/j.apnr.2017.10.004. Epub 2017 Oct 16. PMID 29241512
- [Result] Ferguson RJ, Palmer AJ, Taylor A, Porter ML, Malchau H, Glyn-Jones S. Hip replacement. Lancet. 2018 Nov 3;392(10158):1662-1671. doi: 10.1016/S0140-6736(18)31777-X. PMID 30496081
- [Result] Shin HR, Park K, Seo J, An SH, Yeom SR, Kwon YD. Acupuncture for perioperative care of total hip arthroplasty: A systemic review of controlled trials and meta-analysis. Medicine (Baltimore). 2019 Apr;98(15):e15198. doi: 10.1097/MD.0000000000015198. PMID 30985714
- [Result] OECD, "Hip and knee replacement", in Health at a Glance 2015: OECD Indicators, OECD Publishing, Paris, 2015. doi.org/10.1787/health_glance-2015-36-en
- [Result] Yaban ZŞ, Karaöz S. "Total Kalça Protezi Ameliyatında Hemşirelik Bakımı", C.Ü.Hemşirelik Yüksekokulu Dergisi, 2007; 11 (1):47-53.
- [Result] Widnyana IMG, Senapathi TGA, Aryabiantara IW. "Metabolic Stress Response Attenuate by Oral Glucose Preoperatively in Patient Underwent Major Surgery with General Anesthesia", Int J Anesth Pain Med. 2017; 3(1): 1-5.10.21767/2471-982X.100015
- [Result] Wolf AR. Effects of regional analgesia on stress responses to pediatric surgery. Paediatr Anaesth. 2012 Jan;22(1):19-24. doi: 10.1111/j.1460-9592.2011.03714.x. Epub 2011 Oct 14. PMID 21999144
- [Result] Celiksular MC, Saracoglu A, Yentur E. The Influence of Oral Carbohydrate Solution Intake on Stress Response before Total Hip Replacement Surgery during Epidural and General Anaesthesia. Turk J Anaesthesiol Reanim. 2016 Jun;44(3):117-23. doi: 10.5152/TJAR.2016.65265. Epub 2016 Jun 1. PMID 27366573
- [Result] Jovanovski-Srceva M, Kuzmanovska B, Mojsova M, Kartalov A, Shosholcheva M, Temelkovska-Stevanoska M, Gavrilovska A, Stavridis S, Spirovski Z, Kondov B, Kokareva A, Todorov R, Spirovska T. Insulin Resistance, Glycemia and Cortisol Levels in Surgical Patients who Had Preoperative Caloric Load with Amino Acids. Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2015;36(3):61-70. doi: 10.1515/prilozi-2015-0079. PMID 27442397
- [Result] Juni RP, Duckers HJ, Vanhoutte PM, Virmani R, Moens AL. Oxidative stress and pathological changes after coronary artery interventions. J Am Coll Cardiol. 2013 Apr 9;61(14):1471-81. doi: 10.1016/j.jacc.2012.11.068. PMID 23500310
- [Result] Haga Y, Wada Y, Takeuchi H, Furuya T. Evaluation of modified estimation of physiologic ability and surgical stress in patients undergoing surgery for choledochocystolithiasis. World J Surg. 2014 May;38(5):1177-83. doi: 10.1007/s00268-013-2383-0. PMID 24322176
- [Result] Gül A, Andsoy II, Üstündağ H, Özkaya BÖ, "Assessment of preoperative fasting time in elective general surgery", The Journal of Macro Trends in Health and Medicine, 2013; 1(1): 1-8.
- [Result] Dolgun E, Yavuz M, Eroglu B, Islamoglu A. Investigation of Preoperative Fasting Times in Children. J Perianesth Nurs. 2017 Apr;32(2):121-124. doi: 10.1016/j.jopan.2014.12.005. Epub 2016 Jun 21. PMID 28343637
- [Result] Dolgun E, Taşdemir N, Ter N, Yavuz M. "Cerrahi hastalarının ameliyat öncesi aç kalma sürelerinin incelenmesi", FÜ Sağ. Bil. Tıp Dergisi. 2011; 25(1): 11-15.
- [Result] Soreide E, Eriksson LI, Hirlekar G, Eriksson H, Henneberg SW, Sandin R, Raeder J; (Task Force on Scandinavian Pre-operative Fasting Guidelines, Clinical Practice Committee Scandinavian Society of Anaesthesiology and Intensive Care Medicine). Pre-operative fasting guidelines: an update. Acta Anaesthesiol Scand. 2005 Sep;49(8):1041-7. doi: 10.1111/j.1399-6576.2005.00781.x. PMID 16095440
- [Result] Love C. "Fasting the patient before operation", Journal of Orthopaedic Nursing. 2002;1(6): 41-48.
- [Result] Ludwig RB, Paludo J, Fernandes D, Scherer F. Lesser time of preoperative fasting and early postoperative feeding are safe? Arq Bras Cir Dig. 2013 Jan-Mar;26(1):54-8. doi: 10.1590/s0102-67202013000100012. English, Portuguese. PMID 23702872
- [Result] Brady M, Kinn S, Stuart P. Preoperative fasting for adults to prevent perioperative complications. Cochrane Database Syst Rev. 2003;(4):CD004423. doi: 10.1002/14651858.CD004423. PMID 14584013
- [Result] Pedziwiatr M, Pisarska M, Matlok M, Major P, Kisielewski M, Wierdak M, Natkaniec M, Budzynski P, Rubinkiewicz M, Budzynski R. Randomized Clinical Trial To Compare The Effects Of Preoperative Oral Carbohydrate Loading Versus Placebo On Insulin Resistance And Cortisol Level After Laparoscopic Cholecystectomy. Pol Przegl Chir. 2015 Aug;87(8):402-8. doi: 10.1515/pjs-2015-0079. PMID 26495916
- [Result] Nygren J, Thacker J, Carli F, Fearon KC, Norderval S, Lobo DN, Ljungqvist O, Soop M, Ramirez J; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective rectal/pelvic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):285-305. doi: 10.1007/s00268-012-1787-6. No abstract available. PMID 23052796
- [Result] Kisialeuski M, Pedziwiatr M, Matlok M, Major P, Migaczewski M, Kolodziej D, Zub-Pokrowiecka A, Pisarska M, Budzynski P, Budzynski A. Enhanced recovery after colorectal surgery in elderly patients. Wideochir Inne Tech Maloinwazyjne. 2015 Apr;10(1):30-6. doi: 10.5114/wiitm.2015.48697. Epub 2015 Jan 27. PMID 25960790
- [Result] Tamura T, Yatabe T, Kitagawa H, Yamashita K, Hanazaki K, Yokoyama M. Oral carbohydrate loading with 18% carbohydrate beverage alleviates insulin resistance. Asia Pac J Clin Nutr. 2013;22(1):48-53. doi: 10.6133/apjcn.2013.22.1.20. PMID 23353610
- [Result] Svanfeldt M, Thorell A, Hausel J, Soop M, Rooyackers O, Nygren J, Ljungqvist O. Randomized clinical trial of the effect of preoperative oral carbohydrate treatment on postoperative whole-body protein and glucose kinetics. Br J Surg. 2007 Nov;94(11):1342-50. doi: 10.1002/bjs.5919. PMID 17902094
- [Result] Wang ZG, Wang Q, Wang WJ, Qin HL. Randomized clinical trial to compare the effects of preoperative oral carbohydrate versus placebo on insulin resistance after colorectal surgery. Br J Surg. 2010 Mar;97(3):317-27. doi: 10.1002/bjs.6963. PMID 20101593
- [Result] Yuill KA, Richardson RA, Davidson HI, Garden OJ, Parks RW. The administration of an oral carbohydrate-containing fluid prior to major elective upper-gastrointestinal surgery preserves skeletal muscle mass postoperatively--a randomised clinical trial. Clin Nutr. 2005 Feb;24(1):32-7. doi: 10.1016/j.clnu.2004.06.009. PMID 15681099
- [Result] Amer MA, Smith MD, Herbison GP, Plank LD, McCall JL. Network meta-analysis of the effect of preoperative carbohydrate loading on recovery after elective surgery. Br J Surg. 2017 Feb;104(3):187-197. doi: 10.1002/bjs.10408. Epub 2016 Dec 21. PMID 28000931
- [Result] Smith MD, McCall J, Plank L, Herbison GP, Soop M, Nygren J. Preoperative carbohydrate treatment for enhancing recovery after elective surgery. Cochrane Database Syst Rev. 2014 Aug 14;2014(8):CD009161. doi: 10.1002/14651858.CD009161.pub2. PMID 25121931
- [Result] Hausel J, Nygren J, Lagerkranser M, Hellstrom PM, Hammarqvist F, Almstrom C, Lindh A, Thorell A, Ljungqvist O. A carbohydrate-rich drink reduces preoperative discomfort in elective surgery patients. Anesth Analg. 2001 Nov;93(5):1344-50. doi: 10.1097/00000539-200111000-00063. PMID 11682427
- [Result] Sada F, Krasniqi A, Hamza A, Gecaj-Gashi A, Bicaj B, Kavaja F. A randomized trial of preoperative oral carbohydrates in abdominal surgery. BMC Anesthesiol. 2014 Oct 17;14:93. doi: 10.1186/1471-2253-14-93. eCollection 2014. PMID 25364300
- [Result] Kolcaba K. "Comfort theory and practice: a vision for holistic health care and research", Springer Publishing Co, New York. 2003
- [Result] Wilson L, Kolcaba K. Practical application of comfort theory in the perianesthesia setting. J Perianesth Nurs. 2004 Jun;19(3):164-73; quiz 171-3. doi: 10.1016/j.jopan.2004.03.006. PMID 15195275
- [Result] Yılmaz E, Çeçen D, Toğaç HK, Mutlu S, Kara H, Aslan A. "Ameliyat Sürecindeki Hastaların Konfor Düzeyleri ve Hemşirelik Bakımları", Celal Bayar Üniversitesi Sağlık Bilimleri Enstitüsü Dergisi.2018; 5(1):3-9.
- [Result] Winslow EH, Crenshaw JT. Preoperative fasting. Am J Nurs. 2010 Dec;110(12):12; author reply 12. doi: 10.1097/01.NAJ.0000391216.02330.78. No abstract available. PMID 21107043
- [Result] Abd El-Naby AG, El-Sayed ZM. "Preoperative Fasting Time and Selected Postoperative Outcomes among Patients Undergoing Abdominal Surgeries: Correlation Study", Journal of Health, Medicine and Nursing. 2016; 26:109-119.
- [Result] Demirdağ H, Karaöz S. "Ameliyat öncesi besin/sıvı kısıtlamasına ilişkin hastaların deneyimleri ve hemşirelerin konu ile ilgili bilgi ve uygulamaları", Florence Nightingale Hemşirelik Dergisi. 2015; 23(1): 1-10.
- [Result] Imbelloni LE, Pombo IA, Filho GB. [Reduced fasting time improves comfort and satisfaction of elderly patients undergoing anesthesia for hip fracture]. Rev Bras Anestesiol. 2015 Mar-Apr;65(2):117-23. doi: 10.1016/j.bjan.2013.10.017. Epub 2014 Sep 26. Portuguese. PMID 25740278
- [Derived] Ertural F, Kucukakca Celik G, Ozcelik H. Effect of Oral Carbohydrate Solution Administered Before Hip Arthroplasty on Preoperative Anxiety and Postoperative Patient Comfort: A Randomized Controlled Trial. J Perianesth Nurs. 2023 Jun;38(3):461-468. doi: 10.1016/j.jopan.2022.08.012. Epub 2023 Feb 16. PMID 36803737